CLINICAL TRIAL: NCT00462488
Title: Phase II Study to Evaluate the Efficacy and Tolerability of Intravesical Vicinium™ in Patients With Non-Invasive Urothelial Carcinoma in Situ (CIS) Previously Treated With Bacille Calmette-Guérin (BCG)
Brief Title: Study of Vicinium for Treating Patients With Non-Invasive Urothelial Carcinoma In Situ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sesen Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB4-845-02-IIA
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Urinary Bladder Cancer; Bladder Cancer; Bladder Neoplasms; Bladder Tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — VB4-845

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Schedule A - (Active Comparator): Induction Phase is a single intravesical dose of Vicinium at 30 mg in 40 mL PBS once per week for 6 weeks. If free of disease at 12 weeks after the first instillation, the subject enters Maintenance dosing in which 30 mg of Vicinium is administered once per week for 3 weeks followed by 9 weeks of no therapy.
  If the subject had histologically confirmed disease that is stage <T2, they repeat the Induction phase dosing. If the subject is free of disease, the subject enters the maintenance dosing phase of every 12 weeks (3 weeks of therapy followed by 9 weeks of no therapy until disease recurrence is confirmed by positive biopsy or up to a maximum of Week 51 (end-of-study [EOS]).
  Interventions: Drug: Vicinium
- Treatment Schedule B (Active Comparator): Induction Phase is a single intravesical dose of Vicinium at 30 mg in 40 mL PBS once per week for 12 weeks followed by 1 week of no therapy.
  If 13 weeks after the first instillation of Vicinium the subject is free of disease, they have a break from therapy before entering Maintenance dosing in which 30 mg of Vicinium is administered once weekly for 3 weeks followed by 9 weeks of no therapy. If the subject is free of disease, additional maintenance cycle(s) are repeated every 12 weeks (3 weeks of therapy followed by 9 weeks of no therapy until disease recurrence is confirmed by positive biopsy or up to a maximum of Week 57 (EOS).
  Interventions: Drug: Vicinium

INTERVENTIONS:
Drug: Vicinium — Intravesical administration of Vicinium
  Other Names: VB4-845

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of Vicinium when administered as a monotherapy intravesical instillation in patients with non-invasive urothelial carcinoma in situ (CIS) who failed previous treatment with Bacille Calmette Guérin (BCG).

DETAILED DESCRIPTION:
A phase II study was performed to assess the efficacy and tolerability of intravesical Vicinium in patients with urothelial carcinoma in situ of the bladder. Bacillus Calmette-Guérin treatment had previously failed in all patients. A total of 46 patients were treated with Vicinium with half being administered 30mg/dose once per week for 6 weeks (cohort 1) and the other half (cohort 2) the same dose but administered once per week for 12 consecutive weeks. Disease assessments consisting of urine cytology, cystoscopy and, if indicated, biopsy were performed at 3 month intervals. Patients that were disease-free at the assessment time point were allowed to continue treatment in the maintenance phase which consisted of three weekly doses, followed by 9 weeks of no treatment. As long as the patient remained disease-free, treatment continued for a total of one year.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

* The patient must be male or female 18 years of age or older.
* The patient must have histologically-confirmed Transitional Cell Carcinoma (TCC) of the bladder.
* The patient must have histologically-confirmed carcinoma in situ (CIS), with or without non-invasive papillary disease
* The patient must have immunohistochemically-confirmed EpCAM positive disease.
* The patient must have a life expectancy of at least 12 months.

Prior/Concurrent Therapy

* The patient must have, within the last 24 months, failed to respond to at least 1 cycle of treatment with BCG (with or without interferon) or be intolerant to BCG treatment.
* The patient must have had a transurethral resection of the bladder tumour (TURBT) mapping the location of tumour and quantifying the area of bladder affected.
* The patient must have documented residual CIS (i.e. unresectable disease) prior to study drug administration.

Patient Characteristics

The patient must have adequate organ function, as defined by the clinical trial protocol

Other

* The patient must have the ability to understand and sign an Independent Ethics Committee or Institutional Review Board (IEC/IRB)- approved informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment and is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* The patient has evidence of urethral or upper tract transitional cell carcinoma (TCC) by biopsy or upper tract radiological imaging (i.e. intravenous pyelogram, computed tomography (CT) urogram, or retrograde pyelogram) within the past 2 years
* The patient has hydronephrosis
* The patient has had prior intravesical chemotherapy or investigational or anti-cancer treatments within the last 2 months, inclusive of single-dose adjuvant intravesical chemotherapy immediately post-TURBT
* The patient has existing severe urinary tract infection or recurrent severe bacterial cystitis
* The patient has active, uncontrolled impairment of the renal, hepatobiliary, cardiovascular, gastrointestinal, urogenital, neurologic or hematopoietic systems which, in the opinion of the investigator, would predispose the patient to the development of complications from the administration of intravesical therapy and/or general anesthesia
* Any patient who, in the opinion of the investigator, cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy, biopsy) due to the presence of concomitant serious illness (i.e. uncontrolled cardiac or respiratory disorders)
* The patient is pregnant or breast feeding
* Women of reproductive age (who are not either medically or surgically incapable or bearing children) and all men may not participate unless agreeing to use double barrier contraception, or commit to abstinence during the period of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Chapman, Study Director — Sesen Bio, Inc.
Locations (21):
- United States (8):
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Urology Institute Research, Springfield, Oregon
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Corpus Christi Urology Group, LLP, Corpus Christi, Texas
  - Urology of Virginia, Newport News, Virginia
- Canada (13):
  - Andreou Research, Surrey, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - The Male/Female Health and Research Centre, Royal Court Medical Centre, Barrie, Ontario
  - Urology Resource Centre, Burlington, Ontario
  - McMaster University, Institute of Urology at Saint Joseph's Hospital, Hamilton, Ontario
  - Centre for Applied Urological Research, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario
  - Todd Webster, M.D., Owen Sound, Ontario
  - The Scarborough Hospital, Scarborough Village, Ontario
  - University of Toronto, Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Hopital Fleuimont, Sherbrooke, Quebec

REFERENCES:
- [Derived] Kowalski M, Guindon J, Brazas L, Moore C, Entwistle J, Cizeau J, Jewett MA, MacDonald GC. A phase II study of oportuzumab monatox: an immunotoxin therapy for patients with noninvasive urothelial carcinoma in situ previously treated with bacillus Calmette-Guerin. J Urol. 2012 Nov;188(5):1712-8. doi: 10.1016/j.juro.2012.07.020. Epub 2012 Sep 19. PMID 22998907

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Schedule A -: Induction Phase is a single intravesical dose of Vicinium at 30 mg in 40 mL PBS once per week for 6 weeks. If free of disease at 12 weeks after the first instillation, the subject enters Maintenance dosing in which 30 mg of Vicinium is administered once per week for 3 weeks followed by 9 weeks of no therapy.
  If the subject had histologically confirmed disease that is stage <T2, they repeat the Induction phase dosing. If the subject is free of disease, the subject enters the maintenance dosing phase of every 12 weeks (3 weeks of therapy followed by 9 weeks of no therapy until disease recurrence is confirmed by positive biopsy or up to a maximum of Week 51 (end-of-study [EOS]).
  Vicinium: Intravesical administration of Vicinium
- Treatment Schedule B: Induction Phase is a single intravesical dose of Vicinium at 30 mg in 40 mL PBS once per week for 12 weeks followed by 1 week of no therapy.
  If 13 weeks after the first instillation of Vicinium the subject is free of disease, they have a break from therapy before entering Maintenance dosing in which 30 mg of Vicinium is administered once weekly for 3 weeks followed by 9 weeks of no therapy. If the subject is free of disease, additional maintenance cycle(s) are repeated every 12 weeks (3 weeks of therapy followed by 9 weeks of no therapy until disease recurrence is confirmed by positive biopsy or up to a maximum of Week 57 (EOS).
  Vicinium: Intravesical administration of Vicinium
Period: Overall Study
Arm/Group | Treatment Schedule A - | Treatment Schedule B
Started | 23 | 23
Completed Induction Phase | 22 | 23
Completed Induction 2/Maintenance 1 | 18 | 9
Completed Maintenance 2 | 7 | 6
Completed (Completed the full 51/57 weeks of study) | 3 | 6
Not Completed | 20 | 17
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Schedule A - | Treatment Schedule B | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 18 | 19 | 37
Age, Continuous [Mean (Full Range); unit: years] | 71.6 [41 to 89] | 71.5 [54 to 92] | 71.6 [41 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 17 | 19 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 22 | 22 | 44
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 15 | 30
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Treatment Schedule A: 12-Week Efficacy, Treatment Schedule B: 13-Week Efficacy
Description: Complete response rate in subjects with carcinoma in situ (CIS) non-muscle invasive bladder cancer (NMIBC) following the induction phase (3-month evaluation point) of Vicinium treatment
Time Frame: 12 or 13 weeks
Population: One subject in Treatment Schedule A was not evaluated for complete response after the induction phase as they were ineligible to be on trial and therefore discontinued after receiving one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Schedule A - | Treatment Schedule B
Number analyzed (Participants) | 22 | 23
percentage of patients | 40.9 [20.7 to 63.6] | 39.1 [19.7 to 61.5]

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | Treatment Schedule A - | Treatment Schedule B
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 5/23
Other Adverse Events (participants affected / at risk) | 21/23 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Schedule A - (N=23) | Treatment Schedule B (N=23)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Extravasation during TURBT (Renal and urinary disorders) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Schedule A - (N=23) | Treatment Schedule B (N=23)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 5 (12) | 5 (5)
Influenza like illness (General disorders) | 4 (4) | 2 (4)
Localized Oedema (General disorders) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 3 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4) | 6 (11)
Blood urine present (Investigations) | 2 (2) | 3 (5)
Cells in urine (Investigations) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (10)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2)
Bladder pain (Renal and urinary disorders) | 3 (5) | 2 (3)
Dysuria (Renal and urinary disorders) | 11 (18) | 17 (53)
Haematuria (Renal and urinary disorders) | 8 (16) | 5 (9)
Haemorrhage urinary tract (Renal and urinary disorders) | 2 (2) | 1 (4)
Micturition urgency (Renal and urinary disorders) | 3 (4) | 7 (8)
Nocturia (Renal and urinary disorders) | 2 (2) | 5 (8)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 8 (10)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days